CLINICAL TRIAL: NCT05841511
Title: Effectiveness of Chinese Handwriting Intervention Program for Children With ASD: A Randomized Crossover Trail
Brief Title: Effectiveness of Chinese Handwriting Intervention Program for Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202302086RINB
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: handwriting performance; neurodevelopmental disorder; visual perceptual skills; fine motor skills; visual motor integration skills
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate treatment group (Experimental): The immediate treatment group will receive the intervention in the first time period, while the wait-list control group will receive the intervention program during the second time period. Baseline and outcome evaluation will be accessed at three-time points: baseline assessment (1st week), assessment 1-midway (5th week), and assessment 2-final (10th week) in this study.
  To establish and develop an efficient program, several theories were implemented into the intervention design to address handwriting problems in children with ASD, including psycho-geometric theory, motor learning theory, and cognitive training theories. The intervention will be delivered in thirty-six activities for visual perceptual, fine motor, and visual motor integration skill training integrated with the unique properties of the Chinese writing system. A total of 12 hours of intervention program will be conducted in eight sessions within four weeks.
  Interventions: Behavioral: Chinese handwriting intervention program for children with ASD, named "Go Go Handwriting - ASD version"
- Wait-list control group (Experimental): The immediate treatment group will receive the intervention in the first time period, while the wait-list control group will receive the intervention program during the second time period. Baseline and outcome evaluation will be accessed at three-time points: baseline assessment (1st week), assessment 1-midway (5th week), and assessment 2-final (10th week) in this study.
  To establish and develop an efficient program, several theories were implemented into the intervention design to address handwriting problems in children with ASD, including psycho-geometric theory, motor learning theory, and cognitive training theories. The intervention will be delivered in thirty-six activities for visual perceptual, fine motor, and visual motor integration skill training integrated with the unique properties of the Chinese writing system. A total of 12 hours of intervention program will be conducted in eight sessions within four weeks.
  Interventions: Behavioral: Chinese handwriting intervention program for children with ASD, named "Go Go Handwriting - ASD version"

INTERVENTIONS:
Behavioral: Chinese handwriting intervention program for children with ASD, named "Go Go Handwriting - ASD version" — The intervention program was developed and finalized by a group of occupational therapist specialists in the pediatric field. Thirty-six 20-minute activities with twelve activities for each handwriting fundamental skill were designed in this program.
  All intervention activities were designed based on the characteristic of Chinese characters and included different types of characters.
  The activities designed will also be graded according to the following principle: (1) the similarities between the character given, (2) the complexity of the figure or character in the activities, and (3) the frequency and level of therapist assistance.
  Furthermore, a playful and interesting intervention context will also be integratedinto the program with the design of the adventure journey of an astronaut to further facilitate the motivation and participation of the participants in our program.

SUMMARY:
This research aims to investigate the effectiveness and acceptability of the newly developed Chinese handwriting performance intervention program

ELIGIBILITY:
Inclusion Criteria:

1. first or second grader
2. reported problems with poor handwriting legibility or performed less readable handwriting as claimed by their school teachers or caregivers
3. score at most 33 scores in overall legibility dimension or at-least 45 incorrect strokes in Chinese Handwriting Legibility Assessment for Children (CHLAC)
4. previously diagnosed with ASD
5. and score at least seven scores in Autism Behavior Checklist Taiwan Version (ABC-T) will be included in this study.

Exclusion Criteria:

1. any physical disability affecting the upper limb
2. any hearing or visual impairment
3. intelligence quotient below 70 or previously diagnosed with intellectual disability
4. unable to follow the evaluation instruction.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Changes of Chinese Handwriting Legibility Assessment for Children (CHLAC) | baseline assessment (1st week), assessment 1- midway (5th week), and assessment 2-final (10th week)
  CHLAC is a self-developed assessment tool to measure handwriting legibility. The participants will be requested to copy the printed 10 Chinese characters to 2*2cm squares on the exam sheet. These Chinese characters were selected from three versions of current mandarin textbooks, and those with high-frequency and around-the-average stroke counts were chosen. These chosen characters were then selected to ensure a similar ratio of each character type in the test. A trained examiner will score the character legibility according to handwriting legibility and amounts of incorrect strokes. The handwriting legibility dimensions include size, position, orientation, proportion, and space. The total score for handwriting legibility will be 50, and a higher score indicates more legible handwriting. The incorrect strokes will also be counted; a higher score indicates less legible handwriting.
Changes of The Battery of Chinese Basic Literacy (BCBL) | baseline assessment (1st week), assessment 1- midway (5th week), and assessment 2-final (10th week)
  The BCBL is a standardized assessment to evaluate Chinese reading and writing skills. It consists of reading and writing tests. Only the copying subtest will be administered in this study to measure the handwriting speed of participants. In this test, the participant is requested to correctly and accurately copy 25 Chinese characters printed on the exam sheet (near copy subtest and 25 Chinese characters displayed on a cloth strip (far copy subtest). The number of correct characters written within the prescribed time will be calculated and converted into character copy per minute to represent their handwriting speed.

SECONDARY OUTCOMES:
Changes of Beery-Buktenica Developmental Test of Visual-Motor Integration - Sixth Edition (VMI-6) | baseline assessment (1st week), assessment 1- midway (5th week), and assessment 2-final (10th week)
  Beery-Buktenica Developmental Test of Visual-Motor Integration - Sixth Edition (VMI-6) is a standardized, norm-referenced assessment to measure the integration level between visual and motor systems of an individual using geometric figure copying tasks. Only the full-form test will be administered in our study. The participants were requested to copy the geometric figure printed, and a trained examiner will score the results according to the criteria given in the scoring sheet. A higher score on this test will represent a better visual-motor integration skill.
Changes of Developmental Test of Visual Perception - Third Edition (DTVP-3) | baseline assessment (1st week), assessment 1- midway (5th week), and assessment 2-final (10th week)
  The DTVP-3 is a standardized, norm-reference test used to evaluate the visual perception skills of children between 4 and 12 years old . The test consists of 5 subscales. Only the eye-hand coordination subtest will be assessed in this study to measure the ability of children to integrate the functioning of visual and fine motor control.
Changes of Test of Visual Perceptual Skills - Fourth Edition (TVPS-4) | baseline assessment (1st week), assessment 1- midway (5th week), and assessment 2-final (10th week)
  TVPS-4 is a motor-free visual perception test for individuals between 4 and 18 years of age. There are seven subtests in TVPS-4, including visual discrimination, visual memory, spatial relationships, form constancy, sequential memory, figure-ground and visual closure. The child is requested to choose the correct answer among 4-5 other plausible options based on the instruction, which is different in every subtest. The test was completed when there were five incorrect answers among seven consecutive questions. The raw score can be converted into a scaled score for each subtest, and the sum of the scaled score can be converted into standard scores with a mean of 100 and a standard deviation of 15 to represent the overall test performance. A higher scaled or standard score obtained represents a better visual perception skill.
Changes of Bruininks-Oseretsky Test of Motor Proficiency - Second Edition (BOT-2) | baseline assessment (1st week), assessment 1- midway (5th week), and assessment 2-final (10th week)
  The BOT-2 is a standardized instrument to measure fine motor function in children from 4 to 21 years old. The BOT-2 consists of eight tasks; only two for fine motor control and two for manual coordination will be measured in this study: a fine motor precision task, a fine motor integration task, a manual dexterity, and an upper-limb coordination task. The raw score can be converted into item scaled score and subtest standard score to represent the fine motor performance of the children.
Changes of Pediatric Motivation Questionnaire (PMQ) and Satisfaction Questionnaire for the caregiver (SQ) | baseline assessment (1st week), assessment 1- midway (5th week), and assessment 2-final (10th week)
  Pediatric Motivation Questionnaire (PMQ, Appendix 1) and Satisfaction Questionnaire for the caregiver (SQ, Appendix 2) is our self-developed questionnaire that aims to understand the acceptance of both participants and their caregiver to our program. PMQ and SQ are both five point-Likert scale questionnaires with 12 and 10 questions, respectively. The questions were designed based on three major domains, which include the degree of internal regulation and extrinsic motivation (value or usefulness, effort or importance), basic psychosocial need (relatedness, competence, autonomy), and degree of intrinsic motivation (interest, enjoyment). A higher average score out of 5 indicates the more acceptance and satisfaction with our program.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Department of Occupational Therapy, Taipei, Taiwan